CLINICAL TRIAL: NCT04848805
Title: Liver Transplantation in Patients With Incidental Hepatocellular-cholangiocarcinoma and Intrahepatic Cholangiocarcinoma: A Single-center Experience
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istanbul Demiroglu Bilim University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-243
Record Dates: First submitted 2021-04-02; First posted 2021-04-19 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Adult Combined Hepatocellular-Cholangiocarcinoma
MeSH Terms: interventions — Liver Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- liver recipients with hepatocellular and cohlangiocarcinoma diagnosis: liver recipients
  Interventions: Procedure: liver transplantation

INTERVENTIONS:
Procedure: liver transplantation — total hepatectomy material was examined by pathology laboratory

SUMMARY:
Liver transplantation has become an important treatment in hepatocellular cancer (HCC). While the generally determined malign indication in the world is HCC, some centers perform liver transplantation in both cholangiocarcinoma and mixed type hepatocellular-cholangiocarcinoma diseases and investigate the differences in recurrence and survival outcomes compared to HCC. Although liver transplantation for intrahepatic cholangiocarcinomas of small diameter <2cm is a popular topic of discussion around the world, a common consensus has not been established.

DETAILED DESCRIPTION:
Combined hepatocellular and cholangiocarcinoma (CHC) with an incidence rate from 0.4% to 14.2% in different regions, characterized by hepatocellular and biliary epithelial differentiation within the same tumor, is an unique type of primary hepatic carcinoma that is distinct from hepatocellular carcinoma (HCC) and intrahepatic cholangiocarcinoma (ICC). Combined hepatocellular and cholangiocarcinoma is having attention clinically and pathologically, because of its unique biology, histopathology, and clinical behavior, besides the difficulties in diagnosis and being rare (comprising 1-5% of primary liver cancer). The investigators aimed to present our experience with patients misdiagnosed before LT and found to have incidentally ICC or CHC on explant and compare with HCC, and to identify the demographic, clinical, pathological and etiological risk factors of recurrence and prognostic factors of survival. Liver transplantation has been tried as an effective treatment in mixed-type hepatocellular-cholangiocarcinomas and intrahepatic cholangiocarcinomas, but survival and recurrence-free outcomes have not been achieved as well as HCC. In addition, survival rates reported in different centers also vary. Prognostic factors that may affect disease recurrence and survival include etiology, body mass index, AFP, CEA, CA 19-9, CK7, CK19, CD34, CD56, CD117, CD133, HSA, Arginase, HEPPAR, Amacyr, Glypican 3, Synaptophysin, CK20, CDX2, p53, Ki67, milan criteria, tumor size, tumor number, maximum tumor diameter, total tumor diameter, tumor grade, multicentricity, microvascular invasion, macrovascular invasion, vascular invasion, tumor TNM stage. İnvestigating whether there is a difference between mixed type hepatocellular-cholangiocarcinomas compared to HCC in terms of survival, recurrence and other prognostic markers mentioned above would be important for mixed type tumor relations with liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Explant pathology Being Combined Hepatocellular-Cholangiocarcinoma and Intrahepatic Cholangiocarcinoma
2. Having a liver transplant
3. Being over 18 years old

Exclusion Criteria:

1. Explant pathology being hepatocellular carcinoma
2. Being under the age of 18

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Collected LT database was retrospectively reviewed. 277 patients underwent LT for a primary liver tumor between September 2004 and November 2019 were included in the study. Among these, 17 patients (5%) with incidentally detected CHC and 5 patients (1.8%) with ICCA were included in the study. 257 HCC patients were determined as the control group.
Sampling Method: Probability Sample
Enrollment: 279 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
recurrence | 2005-2020
  correlation between tumor diameter, milan criteria and recurrence

CONTACTS AND LOCATIONS:
Locations (1):
- Group Florence Nightingale Hospitals, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No plan